CLINICAL TRIAL: NCT04853225
Title: Investigation of the Clinical, Radiological and Biological Factors Associated With Disease Progression, Phenotypes and Endotypes of COPD in China
Brief Title: Investigation of Chronic Obstructive Pulmonary Disease (COPD) Phenotypes and Endotypes in China
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Guangzhou Institute of Respiratory Health (GIRH) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 208630
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Phenotypes; Endotypes; Chronic bronchitis; China; Healthy control
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main cohort: COPD, chronic bronchitis and healthy participants (never smoker) from Type A and Type B hospitals will be included.
  Interventions: Other: Prospective observational cohort study
- Sub-cohort: COPD, chronic bronchitis and healthy participants (never smoker) from selected Type A hospitals will be included.
  Interventions: Other: Prospective observational cohort study

INTERVENTIONS:
Other: Prospective observational cohort study — Prospective observational cohort study

SUMMARY:
This is a non-drug interventional cohort study, which aims to investigate the clinical, radiological and biological factors associated with disease progression in COPD in China. Participants will be recruited from multiple hospitals across Guangdong province categorized as Type A hospitals (those at prefecture-level and above) and Type B hospitals (those below prefecture-level).

ELIGIBILITY:
Inclusion criteria:

* Male or female participants, aged 50-80 years inclusive. A female is eligible only if she is of non-child bearing potential.
* Body mass index (BMI) less than (<)35.
* A signed and dated written informed consent is obtained prior to participation.

Additional inclusion criteria for COPD participants:

* A Baseline (post-bronchodilator) (FEV1/FVC) ratio <70 percent (%).
* Clinically stable and has no exacerbations for at least 1 month prior to recruitment.
* Ever smoker or never smoker.

Additional inclusion criteria for chronic bronchitis participants:

* Free from other significant diseases.
* Baseline post-bronchodilator FEV1/FVC ratio more than (>)70%.
* Chronic bronchitis is defined as at least 3 months of cough and phlegm in a year in the past 2 years.
* Clinically stable and has no exacerbations for at least 1 month prior to recruitment.
* Ever smoker or never smoker

Additional inclusion criteria for healthy participants:

* Free from any significant diseases
* Baseline post-bronchodilator FEV1/FVC ratio >70%.
* A CAT score <10.
* Never smoker. Passive smoker is not eligible.

Exclusion criteria:

* Having undergone lung surgery.
* Known respiratory disorders or significant inflammatory disease other than COPD.
* Serious, uncontrolled disease (including serious psychological disorders)
* Confirmed cancer, unless participants in remission for more than or equal to (>=)5 years.
* Participating or plan to participant in any clinical studies where investigational drugs were tested.
* Unable or unwilling to use required digital devices (sub- cohort only).
* Have evidence of alcohol or drug abuse.
* Have received a blood transfusion in the 4 weeks prior to study start.
* On long-term oral corticosteroids.
* Unable to walk.
* Unable to read and understand Mandarin Chinese.

Additional exclusion criteria for COPD participants:

* Current primary diagnosis of asthma (participants with a primary diagnosis of COPD but who also had asthma [Asthma COPD overlap {ACO}] could be included).
* Known disorders other than COPD that may significantly impact clinical assessments

Additional exclusion criteria for chronic bronchitis participants and healthy participants:

* Known disorders that may significantly impact clinical assessments.
* FVC <80% Predicted.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with COPD, chronic bronchitis without fixed airflow limitation and never smoker healthy participants will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2005 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- China (20):
  - GSK Investigational Site, Dongguan
  - GSK Investigational Site, Foshan
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Heyuan
  - GSK Investigational Site, Huizhou
  - GSK Investigational Site, Jiangmen
  - GSK Investigational Site, Jieyang
  - GSK Investigational Site, Meizhou
  - GSK Investigational Site, Qingyuan
  - GSK Investigational Site, Shantou
  - GSK Investigational Site, Shaoguan
  - GSK Investigational Site, Shenzhen
  - GSK Investigational Site, Shunde
  - GSK Investigational Site, Wengyuan
  - GSK Investigational Site, Xiamen
  - GSK Investigational Site, Yunfu
  - GSK Investigational Site, Zhangshan
  - GSK Investigational Site, Zhanjiang
  - GSK Investigational Site, Zhaoqing
  - GSK Investigational Site, Zhuhai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Wen F, Ma Q, Chen R, Sun Y, Liu T, Gu C, Hu S, Song J, Compton C, Zheng J, Zhong N, Jones P. Use of CAPTURE to Identify Individuals Who May or May Not Require Treatment for Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2023 Aug 15;208(4):435-441. doi: 10.1164/rccm.202303-0504OC. PMID 37315325

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2005 participants were enrolled in this study, however only 2003 participants (1 participant withdrew consent and 1 participant withdrew due to investigator discretion) attended Visit 1 creating the Full Population.
Groups:
- COPD Participants: Participants with chronic obstructive pulmonary disease (COPD) were enrolled in this cohort. No study treatment was administered during conduct of this non-interventional study.
- Participants With Chronic Bronchitis: Participants with chronic bronchitis were enrolled in this cohort. No study treatment was administered during conduct of this non-interventional study.
- Never Smoker Healthy Control: Never smoker healthy participants were enrolled in this control cohort. No study treatment was administered during conduct of this non-interventional study.
Period: Overall Study
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Started (Enrolled) | 1698 | 184 | 123
Full Population | 1696 | 184 | 123
Completed | 1451 | 165 | 116
Not Completed | 247 | 19 | 7
Not completed — Withdrawal by Subject | 81 | 4 | 1
Not completed — Physician Decision | 12 | 4 | 1
Not completed — Lost to Follow-up | 50 | 0 | 0
Not completed — Other | 102 | 11 | 5
Not completed — Not included in the Full Population due to Investigator discretion | 1 | 0 | 0
Not completed — Not included in the Full Population due to withdrew consent | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristic data are reported for the Full Population which consisted of all participants who were enrolled in the study and attended Visit 1 (Day 1 of Month 1).
Groups:
- Total: Total of all reporting groups
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control | Total
Number analyzed (Participants) | 1696 | 184 | 123 | 2003
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (7.46) | 61.3 (7.16) | 58.7 (6.72) | 64.6 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 24 | 82 | 282
  Male | 1520 | 160 | 41 | 1721
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 1696 | 184 | 123 | 2003

OUTCOME MEASURES:

1. Secondary Outcome: Main Cohort: Rate of Moderate/Severe Exacerbations in COPD and Chronic Bronchitis Cohorts
Description: Moderate exacerbations are defined as COPD exacerbations that require either systemic corticosteroids (intramuscular, intravenous, or oral) and/or antibiotics. Severe exacerbations are defined as COPD exacerbations requiring hospitalization (including intubation and admittance to an intensive care unit) or result in death. Exacerbation rate = number of moderate or sever exacerbation divided by total participants-years. Analysis performed using a generalized linear model assuming a negative binomial distribution with covariates of type of participants (i.e. GOLD I-IV and chronic bronchitis), gender, smoking status, exacerbation history (moderate/severe), site (type of hospital), maintenance therapy (Y/N) and inhaled corticosteroid (ICS) containing (Y/N), Childhood chest disease (Y/N) and biomass fuel exposure (Y/N), age, and with offset logarithm of time on study.
Time Frame: Up to 30 months
Population: Full Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Number (95% Confidence Interval); unit: Exacerbations per participant per year
Groups:
- Participants With COPD - GOLD Grade I: Participants with COPD classified using the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Grade I (mild COPD) were enrolled in this cohort. No study treatment was administered during conduct of this non-interventional study.
- Participants With COPD - GOLD Grade II: Participants with COPD classified using the GOLD Grade II (moderate COPD) were enrolled in this cohort. No study treatment was administered during conduct of this non-interventional study.
- Participants With COPD - GOLD Grade III: Participants with COPD classified using the GOLD Grade III (severe COPD) were enrolled in this cohort. No study treatment was administered during conduct of this non-interventional study.
- Participants With COPD - GOLD Grade IV: Participants with COPD classified using the GOLD Grade IV (very severe COPD) were enrolled in this cohort. No study treatment was administered during conduct of this non-interventional study.
Arm/Group | Participants With COPD - GOLD Grade I | Participants With COPD - GOLD Grade II | Participants With COPD - GOLD Grade III | Participants With COPD - GOLD Grade IV | Participants With Chronic Bronchitis
Number analyzed (Participants) | 438 | 937 | 223 | 98 | 184
Exacerbations per participant per year | 0.08 [0.06 to 0.10] | 0.12 [0.11 to 0.14] | 0.26 [0.21 to 0.33] | 0.35 [0.25 to 0.49] | 0.02 [0.01 to 0.04]

2. Secondary Outcome: Main Cohort: Change From Baseline in COPD Assessment Test (CAT) Score at Month 30
Description: The CAT is a validated 8-items questionnaire developed for use in routine clinical practice to measure the health status of participants with COPD. Participants rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment), higher score indicates greater impairment. A total CAT score was calculated by summing the non-missing scores of the eight items with a scoring range of 0 (no disease impact) to 40 (maximum disease impact). Higher scores indicated greater disease impact. Baseline value was the assessment with a non-missing value at Day 1 of Month 1. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 of Month 1) and at Month 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1437 | 164 | 116
Scores on a scale | -0.9 (5.84) | -2.3 (5.45) | 0.3 (2.46)

3. Secondary Outcome: Main Cohort: Absolute Values of CAT Score at Month 30
Description: The CAT is a validated 8-items questionnaire developed for use in routine clinical practice to measure the health status of participants with COPD. Participants rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment), higher score indicates greater impairment. A total CAT score was calculated by summing the non-missing scores of the eight items with a scoring range of 0 (no disease impact) to 40 (maximum disease impact). Higher scores indicated greater disease impact.
Time Frame: At Month 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1437 | 164 | 116
Scores on a scale | 7.5 (5.33) | 5.7 (4.18) | 1.3 (2.36)

4. Secondary Outcome: Main Cohort: Total Score of COPD Assessment in Primary Care to Identify Undiagnosed Respiratory Disease and Exacerbation Risk (CAPTURE) at Baseline
Description: The CATPURE is a short, five-item questionnaire that can be easily completed by participants and are used to identify individuals who may have undiagnosed, clinically significant COPD. The algorithm is a simple summation of participants responses to each of the five items. For Question 1-4: Score 0 for 'No' and Score 1 for 'Yes'; Question 5: Score 0 for 'None', 1 for 'Once' and 2 for '2 or more'. Total score is ranging from 0 to 6, higher score means higher risk of COPD (0-1 is at low risk, 2-6 is at high risk). Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: At Baseline (Day 1 of Month 1)
Population: Full Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1696 | 184 | 123
Scores on a scale | 2.6 (1.48) | 2.0 (1.37) | 0.3 (0.55)

5. Secondary Outcome: Main Cohort: Total Score of CAPTURE at Month 18
Description: The CATPURE is a short, five-item questionnaire that can be easily completed by participants and are used to identify individuals who may have undiagnosed, clinically significant COPD. The algorithm is a simple summation of participants responses to each of the five items. For Question 1-4: Score 0 for 'No' and Score 1 for 'Yes'; Question 5: Score 0 for 'None', 1 for 'Once' and 2 for '2 or more'. Total score is ranging from 0 to 6, higher score means higher risk of COPD (0-1 is at low risk, 2-6 is at high risk).
Time Frame: At Month 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1524 | 168 | 117
Scores on a scale | 2.5 (1.48) | 1.8 (1.49) | 0.4 (0.69)

6. Secondary Outcome: Main Cohort: Number of Participants With Any Clinically Important Deterioration (CID) Event and Its Components From Baseline to Month 6
Description: CID was defined as decrease of greater than or equal to (>=) 100 milliliter (mL) in post-bronchodilator FEV1 or increase of >=2 units in the CAT, or an occurrence of a moderate/severe exacerbation. CID was derived from three key clinical assessments: 1. moderate/severe exacerbations, 2. worsening of FEV1, and 3. worsening of health status using the CAT questionnaire. Baseline value was the assessment with a non-missing value at Day 1 of Month 1. A participant may have more than one CID components, hence total of participants with individual CID components may not match with participants with 'Any CID' category. Number of participants with any CID event and its components (Exacerbation CID, FEV1 CID and CAT CID) observed from Baseline to Month 6 have been presented.
Time Frame: Baseline (Day 1 of Month 1) to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1618 | 173 | 122
Participants
  Any CID | 897 | 90 | 58
  Exacerbation CID | 153 | 1 | 0
  FEV1 CID | 431 | 55 | 36
  CAT CID | 567 | 53 | 31

7. Secondary Outcome: Main Cohort: Number of Participants With Any CID Event and Its Components From Months 6 to 18
Description: CID was defined as: decrease of greater than or equal to (>=) 100 milliliter (mL) in post-bronchodilator FEV1 or increase of >=2 units in the CAT, or an occurrence of a moderate/severe exacerbation. CID was derived from three key clinical assessments: 1. moderate/severe exacerbations, 2. worsening of FEV1, and 3. worsening of health status using the CAT questionnaire. A participant may have more than one CID components, hence total of participants with individual CID components may not match with participants with 'Any CID' category. Number of participants with any CID event and its components (Exacerbation CID, FEV1 CID and CAT CID) observed from Months 6 to 18 have been presented.
Time Frame: Months 6 to 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1538 | 169 | 117
Participants
  Any CID | 1120 | 97 | 82
  Exacerbation CID | 211 | 0 | 0
  FEV1 CID | 524 | 64 | 42
  CAT CID | 794 | 52 | 60

8. Secondary Outcome: Main Cohort: Number of Participants With Any CID Event and Its Components From Months 18 to 30
Description: CID was defined as: decrease of greater than or equal to (>=) 100 milliliter (mL) in post-bronchodilator FEV1 or increase of >=2 units in the CAT, or an occurrence of a moderate/severe exacerbation. CID was derived from three key clinical assessments: 1. moderate/severe exacerbations, 2. worsening of FEV1, and 3. worsening of health status using the CAT questionnaire. A participant may have more than one CID components, hence total of participants with individual CID components may not match with participants with 'Any CID' category. Number of participants with any CID event and its components (Exacerbation CID, FEV1 CID and CAT CID) observed from Months 18 to 30 have been presented.
Time Frame: Months 18 to 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1452 | 165 | 116
Participants
  Any CID | 1086 | 93 | 68
  Exacerbation CID | 177 | 2 | 0
  FEV1 CID | 594 | 61 | 37
  CAT CID | 771 | 54 | 48

9. Secondary Outcome: Main Cohort: Number of Participants Who Died
Description: Number of participants who died during study have been presented.
Time Frame: Up to 30 months
Population: Full Population.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1696 | 184 | 123
Participants | 41 | 2 | 0

10. Secondary Outcome: Sub-cohort: Change From Baseline in Evaluating Respiratory Symptoms in COPD (E-RS:COPD) Total Scores From Months 1 to 6
Description: E-RS: COPD is a subset of Exacerbations of Chronic pulmonary Disease Tool (EXACT). E-RS: COPD is a tool that consists of 11 items from the 14 item EXACT instrument. The domains include: respiratory symptoms-breathlessness (RS-BRL) comprised of 5 items (2 items scored from 0-4 and 3 items scored from 0-3); RS-cough and sputum (RS-CSP) comprised of 3 items(2 items scored from 0-4 and 1 item scored from 0-3);and RS-chest symptoms (RS-CSY) comprised of 3 items (scored from 0-4). The total score was calculated by taking sum of all individual 11 item scores, which ranges between 0-40 and higher score indicates more severe symptoms. Baseline value was the assessment with a non-missing value at Day 1 of Month 1. The 1 to 6 month E-RS:COPD total score value was derived by calculating the average of E-RS:COPD total scores collected between month 1 and 6. Change from Baseline was calculated by subtracting Baseline value from 1-6 month average total score value.
Time Frame: Baseline (Day 1 of Month 1) and Months 1 to 6
Population: Sub-cohort Population consisted of participants who were enrolled in the Biomarker and Digital sub-cohort and who provided a least one additional sub-cohort assessment. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 245 | 95 | 53
Scores on a scale | 0.697 (3.6181) | -0.018 (2.8032) | 0.020 (1.2256)

11. Secondary Outcome: Sub-cohort: Change From Baseline in E-RS:COPD Total Scores From Months 18 to 24
Description: E-RS: COPD is a subset of Exacerbations of Chronic pulmonary Disease Tool (EXACT). E-RS: COPD is a tool that consists of 11 items from the 14 item EXACT instrument. The domains include: respiratory symptoms-breathlessness (RS-BRL) comprised of 5 items (2 items scored from 0-4 and 3 items scored from 0-3); RS-cough and sputum (RS-CSP) comprised of 3 items(2 items scored from 0-4 and 1 item scored from 0-3);and RS-chest symptoms (RS-CSY) comprised of 3 items (scored from 0-4). The total score was calculated by taking sum of all individual 11 item scores, which ranges between 0-40 and higher score indicates more severe symptoms. Baseline value was the assessment with a non-missing value at Day 1 of Month 1. The 18 to 24 month E-RS:COPD total score value was derived by calculating the average of E-RS:COPD total scores collected between month 18 and 24. Change from Baseline was calculated by subtracting Baseline value from 18-24 month average total score value.
Time Frame: Baseline (Day 1 of Month 1) and Months 18 to 24
Population: Sub-cohort Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 178 | 70 | 41
Scores on a scale | 1.735 (4.6876) | 1.014 (4.3033) | 0.086 (1.3097)

12. Secondary Outcome: Sub-cohort: Number of Participants With Exacerbation of COPD Tool (EXACT) Events From Months 1 to 6
Description: The EXACT is a 14-item daily diary designed to provide a measure of patient-reported symptoms of COPD exacerbation. An EXACT Total Score, ranging from 0 to 100, where higher scores indicate a more severe condition. EXACT events were defined as magnitude of responder for symptomatic events defined as acute, sustained symptomatic worsening of COPD, defined as an increase in EXACT score >=9 points for 3 days or >=12 points for 2 days, above Baseline (Baseline value is average of 7-day period [Day 1 to 7]). Number of participants with EXACT events observed from Months 1 to 6 have been presented.
Time Frame: Months 1 to 6
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 245 | 95 | 53
Participants | 59 | 12 | 1

13. Secondary Outcome: Sub-cohort: Number of Participants With EXACT Events From Months 18 to 24
Description: The EXACT is a 14-item daily diary designed to provide a measure of patient-reported symptoms of COPD exacerbation. An EXACT Total Score, ranging from 0 to 100, where higher scores indicate a more severe condition. EXACT events were defined as magnitude of responder for symptomatic events defined as acute, sustained symptomatic worsening of COPD, defined as an increase in EXACT score >=9 points for 3 days or >=12 points for 2 days, above Baseline (Baseline value is average of 7-day period [Day 1 to 7]). Number of participants with EXACT events observed from Months 18 to 24 have been presented.
Time Frame: Months 18 to 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 178 | 70 | 41
Participants | 55 | 13 | 0

14. Secondary Outcome: Sub-cohort: Absolute Values of Digital Physical Activity at Baseline (Average of Days 1 to 7)
Description: Digital physical activity was evaluated by daily steps as assessed by a wrist band dispensed at Baseline. Participants were required to keep wearing the wrist band. The daily step data was based on the daily average steps (steps per day) for each participant. Baseline value was derived as the average value of first 7 days (Days 1 to 7 at Month 1).
Time Frame: At Baseline (Days 1 to 7 at Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Steps per day
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 211 | 85 | 49
Steps per day | 7986.2 (3433.46) | 8743.2 (3750.53) | 12063.6 (4152.42)

15. Secondary Outcome: Sub-cohort: Absolute Values of Digital Physical Activity at Month 1 (Average of Day 8 to Month 1)
Description: Digital physical activity was evaluated by daily steps as assessed by a wrist band dispensed at Baseline. Participants were required to keep wearing the wrist band. The daily step data was based on the daily average steps (steps per day) for each participant. Month 1 value was derived as the average of daily step data up to 30 days from study Day 8.
Time Frame: Up to 30 days from study Day 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Steps per day
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 220 | 87 | 52
Steps per day | 8461.3 (3750.31) | 9284.5 (4011.25) | 12790.5 (4233.32)

16. Secondary Outcome: Sub-cohort: Absolute Values of Digital Physical Activity at Month 18 (Average of Months 18 to 19)
Description: Digital physical activity was evaluated by daily steps as assessed by a wrist band dispensed at Baseline. Participants were required to keep wearing the wrist band. The daily step data was based on the daily average steps (steps per day) for each participant. Month 18 value was derived as the average of daily step data up to 30 days from Month 18.
Time Frame: Up to 30 days from Month 18 (Months 18 to 19)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Steps per day
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 170 | 63 | 31
Steps per day | 6138.3 (3664.12) | 6454.3 (3207.73) | 7495.4 (4723.39)

17. Secondary Outcome: Main Cohort: Absolute Values of Plasma Fibrinogen at Baseline
Description: Fibrinogen is a protein, specifically a clotting factor (factor I), that is essential for proper blood clot formation. Blood samples were collected to evaluate the amount of fibrinogen. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: At Baseline (Day 1 of Month 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1694 | 183 | 123
Milligram per deciliter | 337.1 (82.59) | 315.8 (89.97) | 304.4 (73.36)

18. Secondary Outcome: Main Cohort: Absolute Values of Plasma Fibrinogen at Month 30
Description: Fibrinogen is a protein, specifically a clotting factor (factor I), that is essential for proper blood clot formation. Blood samples were collected to evaluate the amount of fibrinogen.
Time Frame: At Month 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1273 | 139 | 102
Milligram per deciliter | 341.2 (82.94) | 328.4 (66.10) | 315.9 (63.01)

19. Secondary Outcome: Main Cohort: Absolute Values of C-Reactive Protein at Baseline
Description: Blood samples were collected for the analysis of C-Reactive Protein. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: At Baseline (Day 1 of Month 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1695 | 183 | 122
Milligram per deciliter | 0.2791 (0.68530) | 0.2463 (0.93353) | 0.1654 (0.40848)

20. Secondary Outcome: Main Cohort: Absolute Values of C-Reactive Protein at Month 30
Description: Blood samples were collected for the analysis of C-Reactive Protein.
Time Frame: At Month 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1272 | 139 | 102
Milligram per deciliter | 0.3411 (0.71558) | 0.2734 (0.63660) | 0.1645 (0.20928)

21. Secondary Outcome: Main Cohort: Absolute Values of Eosinophils and Neutrophils at Baseline
Description: Blood samples were collected for the analysis of eosinophils and neutrophils. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: At Baseline (Day 1 of Month 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1693 | 182 | 120
Giga cells per liter
  Eosinophils | 0.231 (0.2084) | 0.199 (0.1711) | 0.109 (0.1006)
  Neutrophils | 4.467 (1.6253) | 4.180 (1.5366) | 3.810 (0.9967)

22. Secondary Outcome: Main Cohort: Absolute Values of Eosinophils and Neutrophils at Month 30
Description: Blood samples were collected for the analysis of eosinophils and neutrophils.
Time Frame: At Month 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1269 | 139 | 102
Giga cells per liter
  Eosinophils | 0.267 (0.2921) | 0.228 (0.2351) | 0.145 (0.1853)
  Neutrophils | 4.516 (1.6207) | 4.198 (1.6725) | 3.667 (1.0537)

23. Secondary Outcome: Main Cohort: Absolute Values of Hemoglobin at Baseline
Description: Blood samples were collected for the analysis of hemoglobin. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: At Baseline (Day 1 of Month 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1693 | 182 | 120
Grams per liter | 142.2 (13.03) | 141.6 (11.90) | 132.7 (15.03)

24. Secondary Outcome: Main Cohort: Absolute Values of Hemoglobin at Months 30
Description: Blood samples were collected for the analysis of hemoglobin.
Time Frame: At Month 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1269 | 139 | 102
Grams per liter | 143.4 (13.50) | 144.3 (12.29) | 135.3 (12.97)

25. Secondary Outcome: Sub-cohort: Absolute Values of Serum Interferon-gamma-inducible Protein -10 (IP-10) and Serum Soluble Receptor for Advanced Glycation End Products (sRAGE) at Baseline
Description: Blood samples were collected at Baseline for the analysis of blood biomarkers serum IP-10 and serum sRAGE. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: At Baseline (Day 1 of Month 1)
Population: Sub-cohort Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 249 | 98 | 52
Picogram per milliliter
  Serum IP-10 | 41.193 (45.1502) | 36.025 (34.8718) | 48.524 (50.1930)
  Serum sRAGE: number analyzed (Participants) | 248 | 97 | 52
  Serum sRAGE | 907.135 (506.1643) | 993.892 (655.1966) | 1101.124 (551.8240)

26. Secondary Outcome: Sub-cohort: Absolute Values of Serum IP-10 and Serum sRAGE at Month 30
Description: Blood samples were collected at Month 30 for the analysis of blood biomarkers serum IP-10 and serum sRAGE.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 188 | 72 | 42
Picogram per milliliter
  Serum IP-10 | 54.435 (83.4309) | 53.711 (51.1595) | 35.103 (20.8046)
  Serum sRAGE | 1046.746 (632.6992) | 1287.528 (905.2041) | 1166.739 (608.9050)

27. Secondary Outcome: Sub-cohort: Absolute Values of Club Cell Protein (CC16) at Baseline
Description: Blood samples were collected for the analysis of blood biomarker CC16. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: At Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 251 | 99 | 52
Nanogram per milliliter | 8.8512 (6.80359) | 9.2704 (7.29006) | 7.8313 (5.76284)

28. Secondary Outcome: Sub-cohort: Absolute Values of CC16 at Month 30
Description: Blood samples were collected for the analysis of blood biomarker CC16.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 188 | 72 | 42
Nanogram per milliliter | 15.2812 (10.90814) | 15.5412 (10.78253) | 14.4739 (8.45046)

29. Secondary Outcome: Sub-cohort: Absolute Values of Glycated Hemoglobin A1c (HbA1c) at Baseline
Description: Blood samples were collected for the analysis of HbA1c. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: At Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in blood
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 251 | 99 | 53
Percentage of HbA1c in blood | 5.68 (0.660) | 5.87 (0.989) | 5.66 (0.901)

30. Secondary Outcome: Sub-cohort: Absolute Values of HbA1c at Month 30
Description: Blood samples were collected for the analysis of HbA1c.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in blood
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 190 | 73 | 42
Percentage of HbA1c in blood | 5.74 (0.754) | 5.99 (1.227) | 5.83 (0.739)

31. Secondary Outcome: Sub-cohort: Sputum Microbiome as Assessed by Molecular Methods
Description: Sputum microbiome evaluation involves extraction of deoxyribonucleic acid from sputum samples and analyzing it to identify the microbial community present in the samples using molecular methods. There were not enough samples for analysis. Consequently, data was not analyzed, and data will never be analyzed for this outcome measure in the future.
Time Frame: Up to 30 months
Population: Sub-cohort Population. There were not enough samples for analysis. Consequently, data was not analyzed, and data will never be analyzed for this outcome measure in the future.
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 0 | 0 | 0

32. Secondary Outcome: Sub-cohort: Absolute Values of Total Cell Count of Sputum Sample at Baseline
Description: Sputum samples were collected from the participants for assessment of total cell count. Baseline value was the assessment with a non-missing value at Day 1 of Month 1. Data was not collected for "Never Smoker Healthy Control" arm as sputum samples were not collected at Baseline visit for healthy control group as per the Protocol.
Time Frame: At Baseline (Day 1 of Month 1)
Population: Sub-cohort Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. Data was not collected for "Never Smoker Healthy Control" arm as sputum samples were not collected at Baseline visit for healthy control group as per the Protocol.
Measure: Mean (Standard Deviation); unit: Cells per milliliter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 52 | 28 | 0
Cells per milliliter | 545.981 (379.7851) | 529.603 (611.6267) |

33. Secondary Outcome: Sub-cohort: Absolute Values of Total Cell Count of Sputum Sample at Month 30
Description: Sputum samples were collected from the participants for assessment of total cell count.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Cells per milliliter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 87 | 35 | 6
Cells per milliliter | 766.888 (1005.4170) | 550.053 (557.1129) | 835.903 (511.9084)

34. Secondary Outcome: Main Cohort: Number of Participants With COPD Medication
Description: Number of participants with COPD medications received have been presented in separate categories. Data was collected in following categories: Naïve, long-acting muscarinic antagonist (LAMA), long-acting beta agonist (LABA), inhaled corticosteroid (ICS)/LABA, LAMA/LABA, Triple (open), and Triple (closed).
Time Frame: Up to 30 months
Population: Full Population. Data was presented for all participants in a single arm and not separated by their health status (COPD, chronic bronchitis and never smoker) as defined in the SAP as this was non-interventional study and it was not an intent to compare data for COPD medication across participants' health status.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants with chronic obstructive pulmonary disease (COPD), chronic bronchitis and never smoker healthy control were enrolled in this cohort. No study treatment was administered during conduct of this non-interventional study.
Arm/Group | All Participants
Number analyzed (Participants) | 2003
Participants
  Naive | 1649
  LAMA | 102
  LABA | 8
  ICS/LABA | 115
  LAMA/LABA | 77
  Triple (open) | 19
  Triple (closed) | 33

35. Secondary Outcome: Main Cohort: Number of Participants With Change From Baseline in Treatment Pattern
Description: Data was collected in following categories: Step-up (the treatment pattern grade become larger than previous visit), Switch (the treatment pattern changed within a same grade (except grade 0), Stable (the treatment pattern remain the same (except grade 0), Step-down (participants receive treatment and the grade goes down compared with the previous visit), Stop/Missing (No treatment record in the period), and Naïve with respect to their treatment received. Baseline value was the assessment with a non-missing value at Day 1 of Month 1. Number of participants with change from Baseline in treatment pattern have been presented.
Time Frame: Baseline (Day 1 of Month 1) and Month 30
Population: Full Population. Data was presented for all participants in a single arm and not separated by their health status (COPD, chronic bronchitis and never smoker) as defined in the SAP as this was non-interventional study and it was not an intent to compare data for treatment patterns across participants' health status.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 2003
Participants
  Step-up | 104
  Switch | 0
  Stable | 32
  Step-down | 10
  Stop/Missing | 309
  Naive | 1548

36. Secondary Outcome: Number of Participants With COPD Related Outpatient Visits
Description: Number of participants with COPD related outpatient visits have been presented.
Time Frame: Up to 30 months
Population: Health Resource Utilization (HRU) is a subset of Full population which consists of participants who used healthcare resources. Due to feasibility issues in capturing data from certain sites via Hospital Information System (HIS), participants enrolled at those sites were not included in the HRU analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1606 | 178 | 119
Participants | 1240 | 50 | 3

37. Secondary Outcome: Number of Participants With Non-COPD Related Outpatient Visits
Description: Number of participants with non-COPD related outpatient visits have been presented.
Time Frame: Up to 30 months
Population: HRU Population.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1606 | 178 | 119
Participants | 0 | 0 | 0

38. Secondary Outcome: Number of Participants With COPD Related Emergency Visits
Description: Number of participants with COPD related emergency visits have been presented.
Time Frame: Up to 30 months
Population: HRU Population.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1606 | 178 | 119
Participants | 185 | 5 | 0

39. Secondary Outcome: Number of Participants With Non-COPD Related Emergency Visits
Description: Number of participants with non-COPD related emergency visits have been presented.
Time Frame: Up to 30 months
Population: HRU Population.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1606 | 178 | 119
Participants | 291 | 32 | 24

40. Secondary Outcome: Number of Participants With COPD Related Hospitalizations Visits
Description: Number of participants with COPD related hospitalizations visits have been presented.
Time Frame: Up to 30 months
Population: HRU Population.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1606 | 178 | 119
Participants | 276 | 6 | 0

41. Secondary Outcome: Number of Participants With Non-COPD Related Hospitalizations Visits
Description: Number of participants with non-COPD related hospitalizations visits have been presented.
Time Frame: Up to 30 months
Population: HRU Population.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 1606 | 178 | 119
Participants | 0 | 0 | 0

42. Secondary Outcome: Direct Medical Costs Associated With COPD Medications During Study Period
Description: Direct medical costs of out-of-pocket payment and basic insurance were included for following items: Hospital, Outpatient, Emergency, Participant check, Participant therapy and Prescribing costs.
Time Frame: Up to 30 months
Population: HRU Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Chinese Yuan
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 816 | 38 | 2
Chinese Yuan
  Out-of-pocket payment: Hospital: number analyzed (Participants) | 32 | 0 | 0
  Out-of-pocket payment: Hospital | 25416.68 (29042.578) |  |
  Basic Insurance: Hospital: number analyzed (Participants) | 246 | 6 | 0
  Basic Insurance: Hospital | 20069.34 (20912.555) | 9637.41 (3660.536) |
  Out-of-pocket payment: Outpatient: number analyzed (Participants) | 816 | 38 | 1
  Out-of-pocket payment: Outpatient | 2088.99 (3896.868) | 1105.52 (1447.270) | 58.00 (NA) — Standard deviation could not be calculated for single participant.
  Basic Insurance: Outpatient: number analyzed (Participants) | 812 | 23 | 2
  Basic Insurance: Outpatient | 5254.15 (5051.381) | 1773.34 (2593.387) | 268.00 (294.156)
  Out-of-pocket payment: Emergency: number analyzed (Participants) | 102 | 3 | 0
  Out-of-pocket payment: Emergency | 962.12 (1354.719) | 430.46 (190.164) |
  Basic Insurance: Emergency: number analyzed (Participants) | 97 | 2 | 0
  Basic Insurance: Emergency | 1016.38 (1054.997) | 102.58 (119.607) |
  Out-of-pocket payment: Participant check: number analyzed (Participants) | 465 | 20 | 1
  Out-of-pocket payment: Participant check | 1138.82 (2936.166) | 543.96 (368.125) | 58.00 (NA) — Standard deviation could not be calculated for single participant.
  Basic Insurance: Participant check: number analyzed (Participants) | 582 | 14 | 1
  Basic Insurance: Participant check | 3447.89 (4982.828) | 2191.53 (2314.739) | 60.00 (NA) — Standard deviation could not be calculated for single participant.
  Out-of-pocket payment: Participant therapy: number analyzed (Participants) | 205 | 7 | 0
  Out-of-pocket payment: Participant therapy | 1177.49 (5938.384) | 68.26 (155.206) |
  Basic Insurance: Participant therapy: number analyzed (Participants) | 394 | 11 | 1
  Basic Insurance: Participant therapy | 3052.55 (5819.362) | 1014.96 (1381.025) | 17.00 (NA) — Standard deviation could not be calculated for single participant.
  Out-of-pocket payment: Prescribing costs: number analyzed (Participants) | 644 | 19 | 0
  Out-of-pocket payment: Prescribing costs | 2468.19 (4715.511) | 1458.08 (1744.227) |
  Basic Insurance: Prescribing costs: number analyzed (Participants) | 809 | 24 | 1
  Basic Insurance: Prescribing costs | 6330.98 (6999.658) | 1747.48 (2348.413) | 459.00 (NA) — Standard deviation could not be calculated for single participant.

43. Secondary Outcome: Sub-cohort: Absolute Values of Airway Wall Area at Baseline
Description: Airway wall area, in ratio, at Baseline is calculated by dividing airway wall area by total airway area, using low-dose high-resolution computed tomography (HRCT) acquired at Baseline. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 243 | 98 | 49
Ratio | 0.630 (0.0408) | 0.623 (0.0335) | 0.631 (0.0321)

44. Secondary Outcome: Sub-cohort: Absolute Values of Airway Wall Area at Month 30
Description: Airway wall area, in ratio, at Month 30 is calculated by dividing airway wall area by total airway area, using low-dose HRCT acquired at Month 30.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 167 | 62 | 39
Ratio | 0.628 (0.0533) | 0.627 (0.0384) | 0.639 (0.0364)

45. Secondary Outcome: Sub-cohort: Average of Airway Major Inner Diameter at Baseline
Description: Average of airway major inner diameter at Baseline is the averaged longest axis of the airway's cross-section in low-dose HRCT acquired at Baseline. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 243 | 98 | 49
Millimeter | 5.505 (0.9841) | 5.619 (0.7687) | 5.301 (0.8259)

46. Secondary Outcome: Sub-cohort: Average of Airway Major Inner Diameter at Month 30
Description: Average of airway major inner diameter at Month 30 is the averaged longest axis of the airway's cross-section in low-dose HRCT acquired at Month 30.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 167 | 62 | 39
Millimeter | 5.371 (0.8963) | 5.536 (0.8258) | 5.128 (1.0098)

47. Secondary Outcome: Sub-cohort: Average of Airway Minor Inner Diameter at Baseline
Description: Average of airway minor inner diameter at Baseline is the averaged shortest axis of the airway's cross-section in low-dose high-resolution Computed Tomography (HRCT) acquired at Baseline. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 243 | 98 | 49
Millimeter | 4.058 (0.6732) | 4.222 (0.6050) | 3.973 (0.5335)

48. Secondary Outcome: Sub-cohort: Average of Airway Minor Inner Diameter at Month 30
Description: Average of airway minor inner diameter at Month 30 is the averaged shortest axis of the airway's cross-section in low-dose HRCT acquired at Month 30.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 167 | 62 | 39
Millimeter | 3.969 (0.6694) | 4.174 (0.6569) | 3.804 (0.5863)

49. Secondary Outcome: Sub-cohort: Total Airway Count at Baseline
Description: Total airway count at Baseline is derived by summing the number of airway segments identified on low-dose HRCT acquired at Baseline. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Airway Segments
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 243 | 98 | 49
Airway Segments | 353.5 (123.77) | 430.9 (144.01) | 352.0 (122.89)

50. Secondary Outcome: Sub-cohort: Total Airway Count at Month 30
Description: Total airway count at Month 30 is derived by summing the number of airway segments identified on low-dose HRCT acquired at Month 30.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Airway Segments
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 167 | 62 | 39
Airway Segments | 425.8 (174.59) | 542.9 (183.86) | 392.9 (193.63)

51. Secondary Outcome: Sub-cohort: Absolute Values of Perimeter of 10 Millimeter (mm) (Pi10) at Baseline
Description: Pi10 at Baseline is a measure of airway wall thickness, which is calculated by the square root of wall area for a theoretical airway with an internal perimeter of 10 millimeter, using low-dose HRCT acquired at Baseline. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 243 | 98 | 49
Millimeter | 3.892 (0.1361) | 3.917 (0.1318) | 3.905 (0.1367)

52. Secondary Outcome: Sub-cohort: Absolute Values of Pi10 at Month 30
Description: Pi10 at Month 30 is a measure of airway wall thickness, which is calculated by the square root of wall area for a theoretical airway with an internal perimeter of 10 millimeter, using low-dose HRCT acquired at Month 30.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 167 | 62 | 39
Millimeter | 3.836 (0.1571) | 3.860 (0.1826) | 3.842 (0.1163)

53. Secondary Outcome: Sub-cohort: Computed Tomography (CT) Attenuation at the 15th Percentile of the Lung CT Histogram (Perc15) in Residual Volume at Baseline
Description: Perc15 in residual volume (RV) at Baseline is the cut-off value, in Hounsfield Unit (HU), below which are distributed the 15 percent of the voxels with the lowest density in low-dose HRCT, acquired at full expiration at Baseline. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hounsfield Unit
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 218 | 96 | 46
Hounsfield Unit | -893.654 (36.9708) | -829.016 (41.3549) | -804.517 (41.8978)

54. Secondary Outcome: Sub-cohort: Perc15 in Residual Volume at Month 30
Description: Perc15 in residual volume (RV) at Month 30 is the cut-off value, in Hounsfield Unit (HU), below which are distributed the 15 percent of the voxels with the lowest density in low-dose HRCT, acquired at full expiration at Month 30.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hounsfield Unit
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 127 | 54 | 29
Hounsfield Unit | -900.234 (35.0697) | -840.501 (36.8535) | -825.538 (40.4339)

55. Secondary Outcome: Sub-cohort: Perc15 in Total Lung Capacity at Baseline
Description: Perc15 in total lung capacity (TLC) at Baseline is the cut-off value, in Hounsfield Unit (HU), below which are distributed the 15 percent of the voxels with the lowest density in low-dose HRCT, acquired at full inspiration at Baseline. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hounsfield Unit
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 243 | 98 | 49
Hounsfield Unit | -929.370 (23.0575) | -903.261 (23.9101) | -885.743 (22.2715)

56. Secondary Outcome: Sub-cohort: Perc15 in Total Lung Capacity at Month 30
Description: Perc15 in total lung capacity (TLC) at Month 30 is the cut-off value, in Hounsfield Unit (HU), below which are distributed the 15 percent of the voxels with the lowest density in low-dose HRCT, acquired at full inspiration at Month 30.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hounsfield Unit
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 167 | 62 | 39
Hounsfield Unit | -933.063 (24.9625) | -908.850 (20.0450) | -878.913 (32.5519)

57. Secondary Outcome: Sub-cohort: Absolute Values of Low Attenuation Area -950 (LAA-950) at Baseline
Description: LAA-950 at Baseline is percentage (%) of voxels with attenuation less than or equal to (<=)-950 Hounsfield Unit (HU), which is associated with the extent of emphysema, computed using low-dose HRCT acquired at Baseline. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % of voxels with attenuation <=-950 HU
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 243 | 98 | 49
% of voxels with attenuation <=-950 HU | 8.378 (8.4787) | 1.707 (2.3429) | 0.295 (0.3556)

58. Secondary Outcome: Sub-cohort: Absolute Values of LAA-950 at Month 30
Description: LAA-950 at Month 30 is percentage (%) of voxels with attenuation <=-950 Hounsfield Unit (HU), which is associated with the extent of emphysema, computed using low-dose HRCT acquired at Month 30.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % of voxels with attenuation <=-950 HU
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 167 | 62 | 39
% of voxels with attenuation <=-950 HU | 9.765 (9.0580) | 1.977 (2.0639) | 0.360 (0.5297)

59. Secondary Outcome: Sub-cohort: Absolute Values of Disease Probability Measure (DPM) to Assess Gas Trapping at Baseline
Description: Percentage of whole lung associated with gas trapping (GT) as measured by DPM at Baseline. DPM uses low-dose HRCT acquired at both full inspiration (total lung capacity [TLC]) and full expiration (residual volume [RV]) for calculating the percentage of lung volume associated with gas trapping. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % of whole lung associated with GT
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 217 | 96 | 46
% of whole lung associated with GT | 44.898 (17.5307) | 28.978 (20.2675) | 24.832 (18.2977)

60. Secondary Outcome: Sub-cohort: Absolute Values of DPM to Assess Gas Trapping at Month 30
Description: Percentage of whole lung associated with gas trapping (GT) as measured by DPM at Week 30. DPM uses low-dose HRCT acquired at both full inspiration (total lung capacity [TLC]) and full expiration (residual volume [RV]) for calculating the percentage of lung volume associated with gas trapping.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % of whole lung associated with GT
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 127 | 54 | 29
% of whole lung associated with GT | 43.210 (14.2281) | 29.414 (16.1524) | 32.157 (20.1380)

61. Secondary Outcome: Sub-cohort: Absolute Values of DPM to Assess Emphysema at Baseline
Description: Percentage of whole lung associated with emphysema as measured by DPM at Baseline. DPM uses low-dose HRCT acquired at both full inspiration (total lung capacity [TLC]) and full expiration (residual volume [RV]) for calculating the percentage of lung volume associated with emphysema. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: %of whole lung associated with emphysema
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 217 | 96 | 46
%of whole lung associated with emphysema | 13.068 (12.2280) | 2.402 (5.3194) | 0.254 (0.5837)

62. Secondary Outcome: Sub-cohort: Absolute Values of DPM to Assess Emphysema at Month 30
Description: Percentage of whole lung associated with emphysema as measured by DPM at Month 30. DPM uses low-dose HRCT acquired at both full inspiration (total lung capacity [TLC]) and full expiration (residual volume [RV]) for calculating the percentage of lung volume associated with emphysema.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: %of whole lung associated with emphysema
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 127 | 54 | 29
%of whole lung associated with emphysema | 15.093 (12.4986) | 2.518 (3.6730) | 0.877 (1.9884)

63. Secondary Outcome: Sub-cohort: Absolute Values of DPM to Assess Normal Tissue at Baseline
Description: Percentage of whole lung associated with normal tissue (NT) as measured by DPM at Baseline. DPM uses low-dose HRCT acquired at both full inspiration (total lung capacity [TLC]) and full expiration (residual volume [RV]) for calculating the percentage of lung volume associated with normal tissue. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % of whole lung associated with NT
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 217 | 96 | 46
% of whole lung associated with NT | 42.035 (20.8647) | 68.620 (21.7128) | 74.914 (18.3597)

64. Secondary Outcome: Sub-cohort: Absolute Values of DPM to Assess Normal Tissue at Month 30
Description: Percentage of whole lung associated with normal tissue (NT) as measured by DPM at Month 30. DPM uses low-dose HRCT acquired at both full inspiration (total lung capacity [TLC]) and full expiration (residual volume [RV]) for calculating the percentage of lung volume associated with normal tissue.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % of whole lung associated with NT
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 127 | 54 | 29
% of whole lung associated with NT | 41.697 (19.2811) | 68.068 (17.7974) | 66.966 (21.3521)

65. Secondary Outcome: Sub-cohort: Air Volume Ratio (RV/TLC) at Baseline
Description: Air volume ratio at Baseline is defined as air volume at full expiration (FE) (residual volume [RV]) divided by air volume at full inspiration (FI) (total lung capacity [TLC]) multiplied by 100 (expressed as percentage), measured using low-dose HRCT acquired at Baseline. Baseline value was the assessment with a non-missing value at Day 1 of Month 1.
Time Frame: Baseline (Day 1 of Month 1)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % of air volume at FI remaining after FE
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 217 | 96 | 46
% of air volume at FI remaining after FE | 62.821 (15.3924) | 48.535 (15.5070) | 45.617 (13.2394)

66. Secondary Outcome: Sub-cohort: Air Volume Ratio (RV/TLC) at Month 30
Description: Air volume ratio at Month 30 is defined as air volume at full expiration (FE) (residual volume [RV]) divided by air volume at full inspiration (FI) (total lung capacity [TLC]) multiplied by 100 (expressed as percentage), measured using low-dose HRCT acquired at Month 30.
Time Frame: At Month 30
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % of air volume at FI remaining after FE
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 127 | 54 | 29
% of air volume at FI remaining after FE | 61.276 (12.9739) | 48.906 (12.0766) | 51.562 (13.4382)

67. Primary Outcome: Main Cohort: Change From Baseline in Pre-bronchodilator and Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Month 30
Description: FEV1 is a measure of lung function and is defined as the volume of air that can be forced out in one second after taking a deep breath. FEV1 was measured electronically by spirometry. Baseline value was the assessment with a non-missing value at Day 1 of Month 1. Change from Baseline was calculated as the value at Month 30 minus the value at Baseline. Change from Baseline in pre- and post-bronchodilator FEV1 was assessed and summarized. Also, yearly rate of change in FEV1 (pre- and post-bronchodilator) was analyzed using random coefficients models.
Time Frame: Baseline (Day 1 of Month 1) and at Month 30
Population: Full Population consisted of all participants who were enrolled in the study and attend Visit 1. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Participants With COPD - GOLD Grade I | Participants With COPD - GOLD Grade II | Participants With COPD - GOLD Grade III | Participants With COPD - GOLD Grade IV | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 302 | 644 | 148 | 44 | 108 | 78
Milliliter
  Pre-bronchodilator: number analyzed (Participants) | 302 | 644 | 146 | 44 | 108 | 78
  Pre-bronchodilator | -158.9 (273.46) | -93.9 (271.65) | -1.2 (226.44) | -17.3 (141.54) | -144.4 (250.50) | -53.6 (222.51)
  Post-bronchodilator: number analyzed (Participants) | 302 | 638 | 148 | 44 | 107 | 78
  Post-bronchodilator | -168.1 (252.93) | -107.4 (250.66) | -34.7 (207.13) | -33.6 (138.98) | -148.2 (229.19) | -77.2 (200.51)
Statistical Analysis 1: Comparison: Participants With COPD - GOLD Grade I; Test type: Other; Adjusted rate of change = -59.46 — Pre-bronchodilator. Adjusted rate of change was analyzed using Random Coefficient Model. The model was fitted with an unstructured variance-covariance matrix
Statistical Analysis 2: Comparison: Participants With COPD - GOLD Grade I; Test type: Other; Adjusted rate of change = -62.73 — Post-bronchodilator. Adjusted rate of change was analyzed using Random Coefficient Model. The model was fitted with an unstructured variance-covariance matrix
Statistical Analysis 3: Comparison: Participants With COPD - GOLD Grade II; Test type: Other; Adjusted rate of change = -48.54 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 4: Comparison: Participants With COPD - GOLD Grade II; Test type: Other; Adjusted rate of change = -50.32 — [estimate comment as in outcome 67, analysis 2]
Statistical Analysis 5: Comparison: Participants With COPD - GOLD Grade III; Test type: Other; Adjusted rate of change = -22.67 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 6: Comparison: Participants With COPD - GOLD Grade III; Test type: Other; Adjusted rate of change = -33.32 — [estimate comment as in outcome 67, analysis 2]
Statistical Analysis 7: Comparison: Participants With COPD - GOLD Grade IV; Test type: Other; Adjusted rate of change = -20.40 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 8: Comparison: Participants With COPD - GOLD Grade IV; Test type: Other; Adjusted rate of change = -31.08 — [estimate comment as in outcome 67, analysis 2]
Statistical Analysis 9: Comparison: Participants With Chronic Bronchitis; Test type: Other; Adjusted rate of change = -64.74 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 10: Comparison: Participants With Chronic Bronchitis; Test type: Other; Adjusted rate of change = -60.26 — [estimate comment as in outcome 67, analysis 2]
Statistical Analysis 11: Comparison: Never Smoker Healthy Control; Test type: Other; Adjusted rate of change = -27.85 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 12: Comparison: Never Smoker Healthy Control; Test type: Other; Adjusted rate of change = -28.65 — [estimate comment as in outcome 67, analysis 2]

68. Primary Outcome: Main Cohort: Change From Baseline in Pre-bronchodilator and Post-bronchodilator Forced Vital Capacity (FVC) at Month 30
Description: FVC is the total amount of air exhaled during FEV test and is a lung function test that is measured during spirometry. Baseline value was the assessment with a non-missing value at Day 1 of Month 1. Change from Baseline was calculated as the value at Month 30 minus the value at Baseline. Change from Baseline in pre- and post-bronchodilator FVC was assessed and summarized. Also, yearly rate of change in FVC (pre- and post-bronchodilator) was analyzed using random coefficients models.
Time Frame: Baseline (Day 1 of Month 1) and at Month 30
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Participants With COPD - GOLD Grade I | Participants With COPD - GOLD Grade II | Participants With COPD - GOLD Grade III | Participants With COPD - GOLD Grade IV | Participants With Chronic Bronchitis | Never Smoker Healthy Control
Number analyzed (Participants) | 302 | 644 | 148 | 44 | 108 | 78
Milliliter
  Pre-bronchodilator: number analyzed (Participants) | 302 | 644 | 146 | 44 | 108 | 78
  Pre-bronchodilator | -229.2 (358.22) | -161.0 (351.83) | -58.6 (402.70) | -27.3 (352.13) | -139.8 (302.96) | -26.4 (264.49)
  Post-bronchodilator: number analyzed (Participants) | 302 | 638 | 148 | 44 | 107 | 78
  Post-bronchodilator | -241.7 (345.52) | -170.5 (332.35) | -115.8 (344.63) | -101.6 (302.39) | -114.0 (273.44) | -81.9 (227.64)
Statistical Analysis 1: Comparison: Participants With COPD - GOLD Grade I; Test type: Other; Adjusted rate of change = -87.47 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 2: Comparison: Participants With COPD - GOLD Grade I; Test type: Other; Adjusted rate of change = -83.25 — [estimate comment as in outcome 67, analysis 2]
Statistical Analysis 3: Comparison: Participants With COPD - GOLD Grade II; Test type: Other; Adjusted rate of change = -77.54 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 4: Comparison: Participants With COPD - GOLD Grade II; Test type: Other; Adjusted rate of change = -77.41 — [estimate comment as in outcome 67, analysis 2]
Statistical Analysis 5: Comparison: Participants With COPD - GOLD Grade III; Test type: Other; Adjusted rate of change = -60.10 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 6: Comparison: Participants With COPD - GOLD Grade III; Test type: Other; Adjusted rate of change = -73.65 — [estimate comment as in outcome 67, analysis 2]
Statistical Analysis 7: Comparison: Participants With COPD - GOLD Grade IV; Test type: Other; Adjusted rate of change = -45.44 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 8: Comparison: Participants With COPD - GOLD Grade IV; Test type: Other; Adjusted rate of change = -79.49 — [estimate comment as in outcome 67, analysis 2]
Statistical Analysis 9: Comparison: Participants With Chronic Bronchitis; Test type: Other; Adjusted rate of change = -74.39 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 10: Comparison: Participants With Chronic Bronchitis; Test type: Other; Adjusted rate of change = -63.04 — [estimate comment as in outcome 67, analysis 2]
Statistical Analysis 11: Comparison: Never Smoker Healthy Control; Test type: Other; Adjusted rate of change = -25.59 — [estimate comment as in outcome 67, analysis 1]
Statistical Analysis 12: Comparison: Never Smoker Healthy Control; Test type: Other; Adjusted rate of change = -38.69 — [estimate comment as in outcome 67, analysis 2]

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected up to approximately 30 months
Description: Serious and non-serious adverse events (SAEs) were not collected during this study as safety was not a study objective per protocol and there was no potential to collect SAEs and non-SAEs related to any GSK product during the conduct of this non-interventional study. Only all-cause mortality was collected for Full Population (N=2003) since 2 participants from Enrolled Population (N=2005) were not included in the Full Population due to withdrew consent/investigator discretion.
Arm/Group | COPD Participants | Participants With Chronic Bronchitis | Never Smoker Healthy Control
All-Cause Mortality (participants affected / at risk) | 41/1696 | 2/184 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT04853225/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT04853225/SAP_001.pdf